CLINICAL TRIAL: NCT03903328
Title: A Preliminary Study of Prevalence of Sarcopenia Among Elderly Living in Care Facilities in Klang Valley, Malaysia
Brief Title: Prevalence of Sarcopenia Among Elderly Living in Care Facilities in Klang Valley, Malaysia
Status: Completed | Type: Observational
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Pramod Divakara Shenoy, MPT, Head of Department of Physiotherapy and Senior Lecturer, Universiti Tunku Abdul Rahman
Other Study IDs: U/SERC/77/2016
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Sarcopenia; Sarcopenic Obesity
Keywords: muscle strength; physical performance; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Body Height; Hand Strength; Walking Speed

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sarcopenia assessment — Sarcopenia assessment by measurement of Skeletal Muscle mass index, hand grip strength and usual gait speed for 5 meter distance, as per the guidelines of Asia Working group for Sarcopenia study, was carried out.
  Other Names: Height and weight measurements; Skeletal muscle mass index; Hand grip strength; Gait speed

SUMMARY:
The primary aim of this study was to investigate the prevalence of age-related progressive decline in muscle mass and strength (Sarcopenia) among Malaysian elderly residing in long-term care facilities. It is a very important condition to study as it is associated with high incidence of fall, hospitalization and mortality.

DETAILED DESCRIPTION:
Over the past few decades, one condition that prominently affects the muscular system, known as sarcopenia, has captured the attention of healthcare experts and researchers. Sarcopenia is a geriatric syndrome characterized by the involuntary, gradual and generalized deterioration of skeletal muscle mass and strength with advancing age. It is to be noted that while sarcopenia is predominantly a syndrome of the elderly, its development may also be observed in various conditions such as disuse, malnutrition and cachexia, all of which are not exclusive only to the elderly. As of now, there are still ongoing research on an international scale with regards to its epidemiology, risk factors, causative factors, adverse clinical complications, prevention and treatment.

Beginning in 1st of October, 2016, Centres for Disease Control and Prevention (CDC) has finally officialised an International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10- CM) code for sarcopenia after its final proposal since April 2015. This establishment has enabled comprehensible clinical guidelines for diagnosis and treatment of sarcopenia, as well as separate reporting and data collection for sarcopenia in the medical community.

In essence, sarcopenia appears to be one of the most important causes of functional impairment, physical disability and loss of independence in older adults and a prevalence study will help to estimate the deleterious effects of this condition on the elderly living in the care facility, who happen to be the less privileged group as compared to their counterparts dwelling in the community.

ELIGIBILITY:
Inclusion Criteria:

* Currently residing in a long-term care facility
* Ability to walk, with or without the use of any walking aid
* Citizen of Malaysia

Exclusion Criteria:

* Inability to stand for height, weight and gait speed assessments
* Presence of cardiac pacemaker
* Presence of artificial limbs / prosthesis / metal implants
* Difficult or dangerous behaviours
* Severe cardiac, pulmonary, or musculoskeletal disorders
* Severe cognitive impairment or any disability that makes communication impossible
* Presence of terminal illness
* Co-morbidities associated with high risk of falls (e.g. Parkinson's disease or CVA) or that may directly influence affect gait speed

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly living in long-term care facilities (Institutionalized elderly) in Klang valley. Only Seven facilities allowing access to the study subjects were studied
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle mass | 10 minutes
  The skeletal muscle mass was measured using a Research grade Segmental BioImpedance Analyser to help derive the skeletal muscle mass index (Appendicular skeletal muscle mass/square of height= kg/m2)
Grip strength | 1 minute to 10 minutes
  Measurement of muscle strength was done using a Jamar hydraulic handheld dynamometer, only one maximal effort was allowed. However, for erroneous performance another attempt was provided after 10 minutes of rest. The measure was recorded in Kgf.
Gait speed | less the 10 minutes on an average
  Usual gait speed was used as a measure of physical performance, where the subject was required to walk along a 5 meter straight path. Time recorded using a stopwatch and speed recorded in meters per second

CONTACTS AND LOCATIONS:
Overall Officials: PRAMOD D SHENOY, MPT, Principal Investigator — Universiti Tunku Abdul Rahman; sook Fan Yap, FRCP (UK), Study Director — Universiti Tunku Abdul Rahman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abizanda P, Navarro JL, Garcia-Tomas MI, Lopez-Jimenez E, Martinez-Sanchez E, Paterna G. Validity and usefulness of hand-held dynamometry for measuring muscle strength in community-dwelling older persons. Arch Gerontol Geriatr. 2012 Jan-Feb;54(1):21-7. doi: 10.1016/j.archger.2011.02.006. Epub 2011 Mar 2. PMID 21371760
- [Background] Abridged Life Tables, Malaysia, 2012-2015. (2015). Department of Statistics Malaysia. Retrieved from: https://www.statistics.gov.my/index.php?r=column/pdfPrev&id=cWxzRWcvMTZrWFp4UStqQmp3MG9QZz09
- [Background] Arai H, Akishita M, Chen LK. Growing research on sarcopenia in Asia. Geriatr Gerontol Int. 2014 Feb;14 Suppl 1:1-7. doi: 10.1111/ggi.12236. No abstract available. PMID 24450555
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Cruz-Jentoft AJ, Landi F, Schneider SM, Zuniga C, Arai H, Boirie Y, Chen LK, Fielding RA, Martin FC, Michel JP, Sieber C, Stout JR, Studenski SA, Vellas B, Woo J, Zamboni M, Cederholm T. Prevalence of and interventions for sarcopenia in ageing adults: a systematic review. Report of the International Sarcopenia Initiative (EWGSOP and IWGS). Age Ageing. 2014 Nov;43(6):748-59. doi: 10.1093/ageing/afu115. Epub 2014 Sep 21. PMID 25241753